CLINICAL TRIAL: NCT00271921
Title: Does Metabolic Syndrome Exist in Anorexia Nervosa?
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: R03 DK66033 (completed); R03DK066033 (NIH)
Record Dates: First submitted 2005-12-29; First posted 2006-01-04 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Anorexia Nervosa; Metabolic Syndrome
Keywords: eating disorders; anorexia nervosa; body fat distribution; metabolic syndrome; visceral adipose tissue
MeSH Terms: conditions — Anorexia Nervosa; Metabolic Syndrome; Feeding and Eating Disorders | interventions — Caloric Restriction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Calorie controlled diet

SUMMARY:
The purpose of this study is to examine whether body fat distribution changes that occur with weight gain in women recovering from anorexia nervosa are transient or persistent, and if they are associated with other features of Metabolic Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of Anorexia Nervosa (except amenorrhea) (restricting or binge eating/purging subtype)
* Female
* Age 18-40
* Medically stable
* Participation in inpatient or daypatient treatment sufficient to restore patient to a BMI of at least 19.5kg/m²

Exclusion Criteria:

* Additional Major Axis I disorder (including substance abuse or dependence
* On daily prescription medication (including oral contraceptives)
* History of suicide attempt or other self-injurious behavior within the previous 6 months
* Significant current or past medical illness,including diabetes mellitus, heart disease
* Indwelling metallic object (e.g., pacemaker,pump), non-removable metal jewelry or recent metallic ink tattoo

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurel Mayer, MD, Principal Investigator — New York State Psychiatric Institute/Columbia University; Henry Ginsberg, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - St. Luke's Roosevelt Hosptial Center, New York, New York
  - New York State Psychiatric Institute/Columbia University, New York, New York

REFERENCES:
- [Derived] Schebendach J, Mayer LE, Devlin MJ, Attia E, Walsh BT. Dietary energy density and diet variety as risk factors for relapse in anorexia nervosa: a replication. Int J Eat Disord. 2012 Jan;45(1):79-84. doi: 10.1002/eat.20922. Epub 2011 Mar 29. PMID 21448937
- [Derived] Bodell LP, Mayer LE. Percent body fat is a risk factor for relapse in anorexia nervosa: a replication study. Int J Eat Disord. 2011 Mar;44(2):118-23. doi: 10.1002/eat.20801. PMID 20127939
- [Derived] Mayer LE, Klein DA, Black E, Attia E, Shen W, Mao X, Shungu DC, Punyanita M, Gallagher D, Wang J, Heymsfield SB, Hirsch J, Ginsberg HN, Walsh BT. Adipose tissue distribution after weight restoration and weight maintenance in women with anorexia nervosa. Am J Clin Nutr. 2009 Nov;90(5):1132-7. doi: 10.3945/ajcn.2009.27820. Epub 2009 Sep 30. PMID 19793856